CLINICAL TRIAL: NCT06366048
Title: A Model Based on Resected Normal Liver Parenchymal Volume（RNLV）to Predict the Risk of Post-Hepatectomy Liver Failure (PHLF)
Brief Title: A Study on Relationship Between Resected Normal Liver Parenchymal Volume（RNLV）and Post-Hepatectomy Liver Failure (PHLF)
Acronym: RNLV
Status: Active, not recruiting | Type: Observational
Sponsor: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yuan-Yuan Wang, a clinical resident of general surgery department, National Natural Science Foundation of China
Other Study IDs: EHBHKY2022-K-025
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Liver Failure
Keywords: resected normal parenchymal volume (RNLV); postoperative hepatectomy liver failure (PHLF); future liver remnant (FLR)
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHLF group: One group was defined as post-operative liver failure accroding to the PHLF definition of 50-50 criteria and ISGLS criteria.
  Interventions: Diagnostic Test: the different definitions of PHLF according to 50-50 criteria and ISGLS criteria
- No PHLF group: One group was defined as no post-operative liver failure accroding to the PHLF definition of 50-50 criteria nor ISGLS criteria.

INTERVENTIONS:
Diagnostic Test: the different definitions of PHLF according to 50-50 criteria and ISGLS criteria — Our study respectively defined the PHLF according to the 50-50 criteria and the ISGLS criteria in literature review.
  Groups: PHLF group

SUMMARY:
The post-hepatotectomy liver failure (PHLF) is still the most worrisome complication of hepatic resection. Surgeons have always been making efforts to preoperatively predict PHLF using kinds of techniques, scoring systems, and variables. The investigators of this study tried to create an individual predictive model based on the variable, resected normal parenchymal volume (RNLV), then assessing the performance and value of the model in clinical practice.

DETAILED DESCRIPTION:
The investigator launched a large sample-size and retrospective study, enrolling more than a thousand consecutive patients diagnosed with hepatocellular carcinoma (HCC) and intracholangiocarcinoma (ICC) underwent hepatotectomy from the investigator's center. The primary aim of study was to identify whether there was strong correlation between RNLV and PHLF, and the second aim was to further build a combination model based on RNLV and evaluate the value of predicting PHLF in clinical practice. The investigators attached same importance to RNLV, compared to future liver remnant, especially for patients with massive tumors and multiple tumors. The investigators hyperthesized that RNLV could be an indicative variable for surgical safety, and help to form a diversifying method to comprehensively assess the risk of PHLF preoperatively.

ELIGIBILITY:
Inclusion criteria:

* selective hepatectomies;
* histologically confirmed as HCC and ICC
* complete and accessible data

Exclusion criteria:

* any history of Associated Liver Partition and Portal vein ligation for Staged hepatectomy (ALPPS)
* any history of portal vein embolism (PVE)
* any history of tumor rupture
* emergency surgery
* pathologically diagnosed with neither HCC nor ICC
* concomitant resection of gastrointestinal organs, spleenectomy or other organs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1133 consecutive patients diagnosed with hepatocellular carcinoma (HCC) and intracholangiocarcinoma underwent hepatectomies.
Sampling Method: Non-Probability Sample
Enrollment: 1133 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Probability of PHLF was predicted with our individual model based on RNLV. | postoperative day 1 to day 30.
  In our center, an increase international normalized ratio greater than 1.15 and concomitant hyperbilirubinemia more than 23μmol/L on or after postoperative day 5 would be defined as PHLF, according to the International Study Group of Liver Surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-yuan Wang, Study Director — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- The Third Affiliated Hospital of Naval Medical University, Shanhai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After we published our study paper, we would like to share IPD attached to our paper as website links.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After our paper published officially. The final time would be end of March 31st,2024.
Access Criteria: Not sure now.

REFERENCES:
- [Background] Ioannou GN, Green P, Kerr KF, Berry K. Models estimating risk of hepatocellular carcinoma in patients with alcohol or NAFLD-related cirrhosis for risk stratification. J Hepatol. 2019 Sep;71(3):523-533. doi: 10.1016/j.jhep.2019.05.008. Epub 2019 May 28. PMID 31145929
- [Background] Xie DY, Ren ZG, Zhou J, Fan J, Gao Q. 2019 Chinese clinical guidelines for the management of hepatocellular carcinoma: updates and insights. Hepatobiliary Surg Nutr. 2020 Aug;9(4):452-463. doi: 10.21037/hbsn-20-480. PMID 32832496
- [Background] Renner P, Schuhbaum J, Kroemer A, Zeman F, Loss M, Lang SA, Geissler EK, Schlitt HJ, Farkas SA. Morbidity of hepatic resection for intermediate and advanced hepatocellular carcinoma. Langenbecks Arch Surg. 2016 Feb;401(1):43-53. doi: 10.1007/s00423-015-1359-y. Epub 2015 Dec 1. PMID 26627084
- [Background] Xie QS, Chen ZX, Zhao YJ, Gu H, Geng XP, Liu FB. Systematic review of outcomes and meta-analysis of risk factors for prognosis after liver resection for hepatocellular carcinoma without cirrhosis. Asian J Surg. 2021 Jan;44(1):36-45. doi: 10.1016/j.asjsur.2020.08.019. Epub 2020 Sep 28. PMID 32988708